CLINICAL TRIAL: NCT00425815
Title: A Placebo-Controlled Trial of Org 24448 (Ampakine) Added to Atypical Antipsychotics in Patients With Schizophrenia
Brief Title: Org 24448 (Ampakine) for Cognitive Deficits in Schizophrenia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated at Sponsor's request.
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of Maryland (Other); Washington University School of Medicine (Other); Massachusetts General Hospital (Other); Nathan Kline Institute for Psychiatric Research (Other); Columbia University (Other); Duke University (Other); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Stephen R. Marder, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TURNS01
Record Dates: First submitted 2007-01-22; First posted 2007-01-23 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Schizophrenia
Keywords: Cognition; Ampakines; Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — 1-(benzofurazan-5-ylcarbonyl)piperidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Org 24448 250 mg (Experimental): Two capsules (one Org 24448 250 mg capsule and one placebo capsule that is identical to the active treatment) will be ingested orally daily for eight weeks.
  Interventions: Drug: Org 24448
- Og 244448 500 mg (Experimental): Two capsules (two Org 24448 250 mg capsules) will be ingested orally daily for eight weeks.
  Interventions: Drug: Org 24448
- Inactive Capsule (Placebo Comparator): Two capsules (two placebo capsules that are identical to the active treatment) will be ingested orally daily for eight weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Org 24448 — Org 24448 is a moderate-potency selective AMPA positive modulator that enhances the glutamate system in the brain.
  Other Names: Ampakine
  Arms: Og 244448 500 mg; Org 24448 250 mg
Other: Placebo — Placebo comparison
  Arms: Inactive Capsule

SUMMARY:
The TURNS is a National Institute of Mental Health (NIMH) funded contract for the evaluation of new compounds for the treatment of cognitive impairments in schizophrenia (HHSN 27820044 1003C; P.I.: Steve Marder, M.D.). Despite advances in the safety, tolerability, and effectiveness of antipsychotic medications for the treatment of schizophrenia, many patients continue to be plagued by impairments in social and work functioning. Persons with schizophrenia commonly show deficits in a number of areas of cognition that include impairments in attention, memory, and executive functioning (the ability and organize one's behavior). Importantly, a large body of literature now shows a link between cognition and community functioning in schizophrenia. It is believed that treatments that improve cognitive deficits may lead to improvements in work and social functioning.

A promising approach to improve the community functioning of patients with schizophrenia is to develop new agents that treat the cognitive deficits of the illness. One type of pharmacological compound that has shown promise at improving cognition is a group of drugs called ampakines. These drugs are believed to improve the activity of a neurotransmitter system in the brain called the glutamate system. Increased activity of this system has been linked to improvements in cognitive functioning. The current study is an eight-week trial comparing two doses of the ampakine drug, Org 24448, that will be added to patients' current atypical antipsychotic medication. One hundred thirty-five patients with schizophrenia, drawn from seven sites, will participate in the study. Cognition will be measured using a variety of paper-and-pencil and computerized measures from the consensus-derived NIMH Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) cognitive battery. Psychiatric symptoms and the ability to perform community-based tasks of daily living will also be measured. Because previous trials with this drug and other similar drugs have detected lasting cognitive benefits, this trial will also repeat clinical assessments four weeks after completion of the study medication.

DETAILED DESCRIPTION:
This study is an eight-week, randomized, placebo-controlled, parallel group, fixed dose trial comparing two doses of the alpha-amino-3-hydroxy-5-methylisoxazole-4-propionic acid (AMPA) receptor positive modulator, Org 24448, added to a stable dose of atypical antipsychotic medication in 135 patients with schizophrenia studied at seven sites. The primary endpoint for this trial is a composite score derived from the MATRICS cognitive battery. Measures of psychiatric symptoms and functioning are secondary endpoints. Because previous trials in animals and humans with this and other AMPA modulators detected persistence of cognitive benefits, this trial will also repeat clinical assessments at follow-up, four weeks after completion of the study medication.

Primary Objective:

1. Compare the effects of an eight-week trial of Org 24448 250 mg BID, 500 mg BID and placebo upon cognitive function as assessed by the MATRICS cognitive battery.

   Secondary Objectives:
2. Compare the effects of an eight-week trial of Org 24448 250 mg BID, 500 mg BID and placebo upon level of functioning as measured by the SCoRS and UPSA.
3. Compare effects of Org 24448 250 mg BID, 500 mg BID and placebo on overall symptoms measured by the BPRS total, psychotic symptoms measured by the BPRS positive symptom items, and negative symptoms measured by the SANS total.
4. Evaluate tolerability of Org 24448 250 mg BID and 500 mg BID compared to placebo measured by the Side Effect Checklist, AIMS, SAS, study completion rates, and frequency of abnormal laboratory values.

   Tertiary Objective:
5. Evaluate persistence of effects on clinical ratings 4 weeks after completion of the 8-week trial.

Methods:

Study Locations: This study will be coordinated by the study PI, Dr. Goff, and the TURNS Treatment Management Unit under the direction of Dr. Buchanan. Patients will be recruited from the Massachusetts General Hospital and Massachusetts Mental Health Center in Boston (Dr. Goff), the Lemuel Shattuck Hospital and Beth Israel Deaconess Medical Center (Dr. Seidman), the Nathan Kline Institute (Drs. Javitt and Nolan), Washington University Medical Center (Drs. Csernansky and Barch), the Maryland Psychiatric Research Center (Drs. Buchanan and Gold), Duke School of Medicine (Drs. McEvoy and Keefe), the University of California at Los Angeles (Drs. Marder and Green) and Columbia University (Drs. Lieberman and Kimhy). The TURNS is a NIMH-funded contract for the evaluation of new compounds for the treatment of cognitive impairments in schizophrenia (HHSN 27820044 1003C; P.I.: Steve Marder, M.D.). Data management will be performed by the Clinical Trials Data Management Unit of the Nathan Kline Institute under the direction of Jim Robinson, M.S., and statistical analysis will be performed by Dr. Robert McMahon of the Maryland Psychiatric Research Center. Org 24448 and matching placebo capsules will be provided by Organon Pharmaceuticals. Laboratory assays will be performed by Quest Diagnostics.

Subjects: Subjects will include 135 inpatients or outpatients with schizophrenia treated for at least 8 weeks with a stable dose of an atypical antipsychotic other than clozapine. Prior to enrollment, it will be determined that the clinician has optimized the dose of the antipsychotic and maintained the medication at a constant dose for at least 4 weeks. Diagnoses will be confirmed using the SCID. Patients will be excluded for significant medical illness, seizure disorder, substance abuse, or inability to provide informed consent. Because our primary hypothesis is that Org 24448 will improve measures of attention and memory, patients must be capable of completing the neuropsychological battery, but no minimum threshold of cognitive impairment is required for inclusion.

Screening: The diagnosis of schizophrenia will be confirmed by a research psychiatrist using a modified version of the Structured Clinical Interview for DSM IV (SCID). The BPRS, SANS, CDRS and SAS will be administered to verify that inclusionary criteria are met. A physical examination, including neurological exam, will be performed and medical history, vital signs (weight, heart rate, oral temperature, sitting and standing blood pressure), and demographic information will be obtained. Laboratory assessments will include standard screening blood tests: electrolytes, creatinine, blood urea nitrogen (BUN), fasting glucose, liver enzymes, T4, calcium, phosphate, magnesium, albumin and complete blood count (CBC) with differential and platelet count. A pregnancy test will be done in all premenopausal women. A routine urinalysis, drug screen, EKG and EEG with hyperventilation and photic stimulation will also be performed. The screening visits will collect all data required to complete inclusionary and exclusionary criteria except for performance on the MATRICS battery and WTAR, which will be administered as a baseline measurement at week 1 of the stabilization phase to minimize practice effects. In addition, subjects must continue to meet inclusionary and exclusionary criteria on baseline symptom ratings which will be performed at the completion of the stabilization phase (stabilization week 2).

Stabilization Phase: After informed consent is obtained and screening completed, subjects will enter a two-week, single-blind placebo lead-in stabilization phase. Placebo will be administered as two capsules twice daily dispensed in blister packs identical to those that will be used during the randomized, double-blind treatment phase. Baseline assessments will be completed during the stabilization phase and compliance with study medication will be assessed. Plasma will be obtained for assay of antipsychotic concentrations at week 2 of the stabilization phase. The plasma sample will be drawn as a trough level. This phase is intended to reduce placebo-response during the double-blind treatment phase, allow completion of baseline assessments, and provide an opportunity for investigators to identify and resolve potential problems with compliance.

The MATRICS Consensus Cognitive Battery (MCCB), the Wechsler Test of Adult Reading (WTAR), the Schizophrenia Cognitive Rating Scale (SCoRS), and the University of California San Diego (UCSD) Performance-Based Skills Assessment (UPSA) will be completed at stabilization week 1; the clinical scales (described under "Assessments") will be completed at stabilization week 2.

Double-Blind Phase: Patients will be randomized in a 1:1:1 ratio to placebo, Org 24448 250 mg BID or Org 24448 500 mg BID administered in identical-appearing capsules for eight weeks. Study drug will be dispensed weekly in blister packs containing placebo or Org 24448 250 mg capsules after completing the stabilization phase (stabilization week 2 and baseline assessments). Subjects will be given three extra days of medication in case of a missed appointment. All subjects will take two capsules twice daily. The antipsychotic dose will be unchanged during the trial. Patients will be asked to bring their previous blister pack to each visit; a count of remaining capsules will be performed and recorded. Patients will return for follow-up at week 12, four weeks after completing the double-blind trial. Investigators may reduce the morning (AM) dose of study drug by one capsule (250 mg) if necessary due to poor tolerance. Subjects may continue at the reduced dose or, after one week, the investigator may attempt to resume the full dose (two capsules BID). If the reduced dose (three capsules daily) is not tolerated, subjects will be discontinued from the study. Patients who miss 7 consecutive days of study drug or who are found to have taken 75% or fewer study doses at two or more pill counts will be dropped from study.

Assessments: The following scales will be completed at stabilization week 2 (baseline) and at weeks 2, 4, 6, 8 & 12 and will comprise the clinical assessment battery: Brief Psychiatric Rating Scale (BPRS), Scale for Assessment of Negative Symptoms (SANS), Calgary Depression Rating Scale (CDRS) and Clinical Global Impression (CGI). In addition, the Abnormal Involuntary Movement Scale (AIMS) and the Simpson Angus Scale for Extrapyramidal Symptoms (SAS) will be performed at baseline and weeks 4, 8 & 12. Assessment of functioning will be performed at baseline, weeks 4 & 8 (or end of study) using the Schizophrenia Cognitive Rating Scale (SCoRS) and UCSD Performance-based Skills Assessment (UPSA). The SCoRS will be repeated at week 12. Cognitive functioning will be assessed at baseline, week 4 and week 8 (or end of study) using the MATRICS battery plus the NAB Daily Living Memory and a Delayed Recall Trial of the Hopkins Verbal Learning Test. A one-week window (up to 3 days before or 4 days after the scheduled visit) will be allowed for the completion of assessments to accommodate unusual or unavoidable circumstances only. All sites will be certified in the administration of the MATRICS, SCoRS and UPSA assessments prior to initiation of study. Inter-rater reliability will be established for the BPRS and SANS before the start of the study and will be reassessed every three months by the circulation of videotaped interviews.

Safety Assessments: Vital signs and the Side Effects Checklist will be performed and adverse events recorded weekly during the two-week stabilization phase and the 8 week trial and weekly for 4 weeks following completion of the trial . Laboratory assessments, including urinalysis, will be repeated at weeks 4, 6 and 8 (or end of study). An EKG will be repeated at weeks 2, 4 and 8. A white blood count (WBC) and absolute neutrophil count (ANC) will be repeated weekly during the 8 week trial and weekly for 4 weeks following completion of the trial. A physical examination, including neurological examination, will be repeated at week 8 (or end of study).Drug Plasma Concentrations: Plasma will be obtained at baseline and weeks 4 and 8 for assay of antipsychotic concentrations. Plasma samples will be drawn as trough levels.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis: schizophrenia, any subtype (DSM-IV/DSM-IV-TR)
2. Age: 18-55 years
3. Gender: male or female
4. Capable of providing informed consent
5. Antipsychotic: aripiprazole, olanzapine, quetiapine, risperidone or ziprasidone.
6. Subjects must have been maintained on current psychotropic medications for 8 weeks and on current doses for 4 weeks.
7. Subjects must be clinically stable and in the residual (non-acute) phase of their illness for at least 12 weeks.
8. Symptom Ratings:

   * No more than a "moderate" severity rating on hallucinations and delusions (i.e., Brief Psychiatric Rating Scale (BPRS) Hallucinatory Behavior or Unusual Thought Content item score 4)
   * No more than a "moderate" severity rating on positive formal thought disorder (i.e., BPRS Conceptual Disorganization item score 4)
   * No more than "moderate" severity rating on negative symptoms (i.e., all Scale for the Assessment of Negative Symptoms global items 3)
   * A minimal level of extrapyramidal symptoms (i.e., Simpson-Angus Scale total score 6)
   * A minimal level of depressive symptoms (i.e., Calgary Depression Scale total score 10).
9. Cognitive Status:

   * Performance less than the maximum cutoff (in parentheses) for ONE of the following MCCB tests:
   * Letter-number span (.20)
   * Hopkins Verbal Learning Test (HVLT) total (.31) and
   * Continuous Performance Test- Identical Pairs (CPT) d-prime (.3.47)
   * Able to complete the baseline MCCB validly as assessed by Chief Neuropsychologist or neuropsychology tester
   * Raw score of 6 or greater on the WTAR

Exclusion Criteria:

1. Concomitant medications are allowed except for:

   * Conventional antipsychotics and clozapine
   * Antipsychotic polypharmacy
   * Anticholinergic agents (including anticholinergic antidepressants)
   * Carbamazepine, phenytoin and lamotrigine
2. DSM-IV/DSM-IV-TR diagnosis of alcohol or substance abuse (other than nicotine) within the last 3 months or a DSM-IV/DSM-IV-TR diagnosis of alcohol or substance dependence (other than nicotine) within the last 6 months
3. A history of significant head injury/trauma, as defined by:

   * Loss of consciousness (LOC) for more than 1 hour
   * Recurring seizures resulting from the head injury
   * Clear cognitive sequelae of the injury
   * Cognitive rehabilitation following the injury
4. History of seizures or abnormal EEG
5. Epileptogenic abnormalities on screening EEG
6. A baseline white blood count (WBC) less than 3500/mm3 or absolute neutrophil count (ANC) less than 2000/mm3
7. Serious medical or neurological illness (unstable cardiac disease, AIDS, malignancy, liver or renal impairment) or treatment for a medical disorder that could interfere with study participation.
8. History of transient ischemic attack (TIA) or cerebral vascular accident (CVA)
9. History of neutropenia or medication-induced blood dyscrasia
10. Clinically-significant abnormalities on screening laboratory or EKG.
11. Untreated hyper- or hypothyroidism
12. Pregnancy, nursing, or if female and fertile, unwilling to use appropriate birth control measures during study participation
13. Unable to complete neuropsychological tests
14. Serious suicidal or homicidal risk within the past six months
15. Participation in a trial of another investigational agent within 2 months
16. Treatment with Electroconvulsive therapy (ECT) within 2 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
MCCB: MATRICS Consensus Cognitive Battery | Baseline, Week 4 and Week 8
  The MATRICS Consensus Cognitive Battery assesses cognitive function in the following domains: speed of processing, attention/vigilance, verbal learning, visual learning, reasoning and problem solving, and social cognition.

SECONDARY OUTCOMES:
UPSA: UCSD Performance-Based Skills Assessment | Baseline, Week 4 and Week 8
  The UPSA assesses skills necessary for functioning in the community by asking patients to perform relevant tasks, rating their performance in five areas: household chores, communication, finance, transportation, and planning recreational activities.
SCoRS: Schizophrenia Cognition Rating Scale | Baseline, Week 4 and Week 8
  The SCoRS is an assessment of cognitive deficits and the degree to which they affect day-to-day functioning. The items assess the cognitive domains of attention, memory, reasoning and problem solving, working memory, processing speed, language functions, and social cognition.

CONTACTS AND LOCATIONS:
Overall Officials: Don C Goff, MD, Principal Investigator — Harvard University
Locations (8):
- United States (8):
  - UCLA, Los Angeles, California
  - Maryland Psychiatric Research Center, Catonsville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Harvard Medical School, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Nathan Kline Institute, Orangeburg, New York
  - Duke University Medical Center, Durham, North Carolina